CLINICAL TRIAL: NCT04943302
Title: Isatuximab and Bendamustine in Systemic Light Chain Amyloidosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left institution. Study not moving forward in her absence.
Sponsor: Tufts Medical Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 00001665
Record Dates: First submitted 2021-06-23; First posted 2021-06-29 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Amyloidosis; Light Chain (AL) Amyloidosis
Keywords: isatuximab; bendamustine
MeSH Terms: conditions — Amyloidosis | interventions — Bendamustine Hydrochloride; isatuximab

STUDY DESIGN:
Intervention Model Description: Phase II, non-randomized, single institution study using a two-stage Simon optimal design. There will first be a safety run-in of 6 patients who will be evaluated for toxicity in cycle 1. Unexpected toxicities will trigger an early safety interim analysis to ensure the regimen is tolerable. In the first stage, 19 patients, including the 6 patients in the safety run-in, will be accrued. If 6 or fewer of these 19 patients achieves hematologic PR, the study will be stopped. Otherwise, up to 20 additional patients will be accrued for a maximum of 39 patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Isatuximab + bendamustine (Experimental): Bendamustine will be administered by IV at a dose of 70mg/m2 on cycle days 1 and 8 for up to 6 cycles. Isatuximab will be administered by IV at a dose of 10mg/kg on cycle 1 days 1, 8, 15, and 22; cycle 2-6 days 1,8; and cycle 7-12 day 1.
  Interventions: Drug: Bendamustine Hydrochloride; Drug: Isatuximab

INTERVENTIONS:
Drug: Bendamustine Hydrochloride — To be given by IV at 70mg/m2 on cycle days 1 and 8 for up to 6 cycles
Drug: Isatuximab — To be given by IV at10mg/kg IV on cycle 1 days 1,8,15, and 22; cycle 2-6 days 1,8; and cycle 7-12 days 1

SUMMARY:
Patients with systemic light chain (AL) amyloidosis, particularly those who are ineligible for transplant or have relapsed/refractory disease, have limited treatment options. The combination of bendamustine and dexamethasone is well-tolerated and efficacious in patients with relapsed/refractory AL amyloidosis. Anti-CD38 antibodies have recently demonstrated great efficacy in AL amyloidosis. Adding isatuximab, a monoclonal antibody targeting CD38, to bendamustine would combine two mechanisms of targeting the clonal plasma cell without significant overlap in toxicity. This would provide a steroid minimizing and neurotoxic-free regimen for patients with AL amyloidosis. This study is a phase II clinical trial of isatuximab and bendamustine in newly diagnosed or relapsed/refractory AL amyloidosis. It is hypothesized that this combination will result in a high number of deep hematologic responses.

DETAILED DESCRIPTION:
Systemic light-chain amyloidosis is a disorder in which clonal plasma cells produce misfolded immunoglobulin light chains that deposit in tissues resulting in organ dysfunction and ultimately death. The incidence in the United States is estimated to be 9.7 to 14.0 cases per million person-years with median survival from diagnosis between 6 months and 3 years.

The standard of care for those who are eligible is high dose chemotherapy with ASCT. However, only 20-25% of patients are eligible for ASCT with another one-third of patients becoming eligible after bortezomib-based induction. Transplant ineligible patients and patients with relapsed disease after transplant are treated with evolving combinations of anti-plasma cell agents adapted from multiple myeloma including melphalan, cyclophosphamide, proteasome inhibitors, immunomodulatory agents with no therapies approved specifically for this disease.

Bendamustine is an alkylating agent that has established anti plasma cell efficacy in both first-line and refractory multiple myeloma. Known for its efficacy and tolerability in a wide array of hematologic malignancies, toxicity profile consists of cytopenias, gastrointestinal side effects, and allergic reactions. In patients with indolent non-Hodgkin's lymphoma, bendamustine with rituximab showed superior 5 year event free survival compared to R-CHOP or R-CVP with a more tolerable toxicity profile.

The tolerability of bendamustine made it an attractive agent for AL amyloidosis given the older patient population and co-existence of organ impairment. Efficacy of bendamustine in AL amyloidosis was recently demonstrated in a multicenter phase II study of 31 patients with relapsed/refractory AL amyloidosis who were given bendamustine 100mg/m2 on days 1 and 2 and dexamethasone 40mg weekly of 28 day cycle (2-12 cycles, median 4 cycles). Hematologic response of very good partial response (VGPR) or greater was achieved in 29% of patients (11% complete response) at median of 2.8 months and 29% achieved organ response. The median overall survival (OS) was 18.2 months, but the median OS was not reached among patients who achieved a hematologic partial response (PR) or better after 2 cycles at a median follow up of 14.9 months. Overall, treatment was well tolerated; the most common grade 3/4 toxicities were leukopenia, fatigue, renal dysfunction, rash, and mood symptoms.

Plasma cells are known to express CD38, including the monoclonal plasma cells that result in AL amyloidosis. Monoclonal antibodies targeting CD38 have become standard of care in multiple myeloma and more recently have demonstrated safety and superior efficacy when combined with cyclophosphamide, bortezomib, and dexamethasone (CyBorD) compared to CyBorD alone in patients with newly diagnosed AL amyloidosis.

Isatuximab is a monoclonal antibody that binds CD38 expressed on plasma cells and results in toxicity and lysis of the cell. Efficacy has been demonstrated in relapsed/refractory multiple myeloma based on a randomized, multicenter, phase 3 clinical trial comparing isatuximab, pomalidomide, and dexamethasone to pomalidomide and dexamethasone which resulted in a significant improvement in PFS (11.5 months vs. 6.5 months; HR 0.596; p=0.001). An ongoing trial, S1702, is investigating isatuximab in patients with relapsed or refractory AL amyloidosis (NCT03499808).

This study proposes the combination of isatuximab and bendamustine as a neurotoxic-sparing and steroid-minimizing regimen for newly diagnosed or relapsed/refractory AL amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Histopathologically confirmed AL amyloidosis based on detection by polarizing microscopy of green birefringent material in Congo Red stained tissue specimens or characteristic electron microscopy appearance or immunohistohemical stain with anti-light chain anti-sera. Diagnosis cannot be based solely on congo red stain on bone marrow biopsy.
3. Measurable disease (one of the following):

   1. Serum monoclonal protein ≥ 0.5g/dL
   2. Urine monoclonal protein >200mg/dL in 24 hour urine collection
   3. Clonal population of plasma cells in the bone marrow
   4. dFLC > 40mg/L
4. Mayo Cardiac Amyloid Stage I-IIIA based on the Mayo 2004/European Addition criteria
5. ECOG 0-2
6. ANC ≥ 1.0 x10^9/L
7. Hemoglobin ≥ 8g/dL
8. Platelet count ≥ 75 x10^9/L
9. Calculated creatinine clearance ≥ 30mL/min based on the Cockcroft-Gault formula
10. AST and ALT ≤ 2.5x ULN
11. Serum bilirubin < 1.5x ULN
12. Willingness to provide consent and participate in study activities
13. Male participants must agree to use contraception during the intervention period and for at least 5 months after the last dose of isatuximab treatment and refrain from donating sperm during this period.
14. Female participants may not be pregnant, not be breastfeeding, and at least one of the following conditions apply:

    1. Not a female of childbearing potential
    2. A female of childbearing potential who has a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours prior to starting study medication and before each cycle of study treatment and must either commit to continue abstinence from heterosexual intercourse or apply a highly effective method of birth control during the intervention period and for at least 5 months after the last dose of isatuximab treatment

Exclusion Criteria:

1. Resistant to prior anti CD38 antibody therapy as defined as either non-responsive or progression while on or within 60 days of discontinuation of treatment
2. Received anti CD38 antibody in the previous 6 months
3. Active symptomatic multiple myeloma as defined by IMWG. Smoldering multiple myeloma is permissible.
4. Myocardial infarction within 6 months prior to enrollment.
5. NYHA class IIIB or IV heart failure
6. Mayo Cardiac Amyloid Stage IIIB based on the Mayo 2004/European Addition criteria (See Appendix A)
7. Uncontrolled angina
8. Severe uncontrolled ventricular arrhythmias
9. Active conduction system abnormalities not including 1st degree AV-block, Wenckebach type 2nd degree heart block, or left bundle branch block.
10. Use of other investigational drug within 14 days or 5 half-lives of the investigational drug prior to initiation of study intervention, whichever is longer.
11. Any clinically significant, uncontrolled medical condition that, in the investigator's opinion, would expose the patient to excessive risk or may interfere with compliance or interpretation of the study results.
12. Active systemic infection and severe infections requiring treatment with parenteral administration of antibiotics.
13. Known to be HIV+ or to have hepatitis A, B, or C active infection

    1. Uncontrolled or active HBV infection: Patients with positive HBsAg and/or HBV DNA

       * Patients can be eligible if anti-HBc IgG positive (with or without positive antiHBs) but HBsAg and HBV DNA are negative.
       * If anti-HBV therapy in relation with prior infection was started before initiation of IMP, the anti-HBV therapy and monitoring should continue throughout the study treatment period.
       * Patients with negative HBsAg and positive HBV DNA observed during screening period will be evaluated by a specialist for start of anti-viral treatment: study treatment could be proposed if HBV DNA becomes negative and all the other study criteria are still met.
    2. Active HCV infection: positive HCV RNA and negative anti HCV

       * Patients with antiviral therapy for HCV started before initiation of IMP and positive HCV antibodies are eligible. The antiviral therapy for HCV should continue throughout the treatment period until seroconversion.
       * Patients with positive anti-HCV and undetectable HCV RNA without antiviral therapy for HCV are eligible.
14. Pregnancy or breastfeeding
15. Treatment or diagnosis of another malignancy within 3 years of enrollment except complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, low risk prostate cancer.
16. Hypersensitivity to bendamustine
17. Hypersensitivity or history of intolerance to steroids, mannitol, pregelatinized starch, sodium stearyl fumarate, histidine (as base and hydrochloride salt), arginine hydrochloride, poloxamer 188, sucrose or any of the other components of study intervention that are not amenable to premedication with steroids and H2 blockers or would prohibit further treatment with these agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Estimated Hematologic Response | 36 Months
  Hematologic complete response + very good partial response (CR+VGPR) with definitions as follows:
  * CR: Normalization of free light chain (FLC) ratio AND negative serum and urine immunofixation
  * VGPR: Reduction in the difference between involved and uninvolved free light chains (dFLC) to <40mg/L
  * Partial response (PR): Reduction in the dFLC to at least 50%
  * No response (NR): Less than a PR

SECONDARY OUTCOMES:
Organ Response Rate | 36 Months
  Organ response rate as defined by:
  * Kidneys: 30% reduction in 24-hour urine protein excretion or a drop of proteinuria below 0.5g/24h in the absence of progressive renal insufficiency, defined as a decrease in eGFR to 25% over baseline.
  * Heart: Reduction of NT-proBNP of 30% and >300ng/L decrease from the starting value with baseline NT-proBNP ≥650ng/L OR reduction of BNP of 30% and >50ng/L from the starting value with baseline BNP ≥150ng/L.
  * Liver: 50% decrease of an initially elevated alkaline phosphatase level or reduction in the size of the liver by at least 2cm (determined by physical exam, ultrasound, or computer tomography)
  * Neuropathy: clinical improvement supported by clinical history, neurologic exam, orthostatic vital signs, resolution of severe constipation or reduction of diarrhea to less than 50% of previous movements/day, and EMG studies if indicated
Progression-Free Survival (PFS) | 36 Months
  PFS per the IMWG definition of progression of disease:
  * From CR: Any detectable monoclonal protein or abnormal free light chain ratio (involved light chain must double)
  * From PR: 50% increase in serum M protein to >0.5g/dL or 50% increase in urine M protein to >200mg/day (a visible peak must be present)
  * Free light chain increase of 50% to >100mg/L
Rates if Bone Marrow MRD | 36 Months
  Bone marrow MRD negativity by NGS at a sensitivity of 1x10-6 at the time of complete response, end of treatment visit, and end of study visit.
Time to Next Treatment | 36 Months
  Time to next treatment
Toxicity of the Regimen | 36 Months
  Toxicity assessment with CTCAE v5.0
Peripheral Blood BCMA Levels (exploratory) | 36 Months
  Peripheral blood BCMA levels as assayed by the Comenzo Laboratory at Tufts Medical Center.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Varga, MD, Principal Investigator — Tufts Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gertz MA. Immunoglobulin light chain amyloidosis: 2020 update on diagnosis, prognosis, and treatment. Am J Hematol. 2020 Jul;95(7):848-860. doi: 10.1002/ajh.25819. Epub 2020 Apr 28. PMID 32267020
- [Background] Quock TP, Yan T, Chang E, Guthrie S, Broder MS. Epidemiology of AL amyloidosis: a real-world study using US claims data. Blood Adv. 2018 May 22;2(10):1046-1053. doi: 10.1182/bloodadvances.2018016402. PMID 29748430
- [Background] Cornell RF, Zhong X, Arce-Lara C, Atallah E, Blust L, Drobyski WR, Fenske TS, Pasquini MC, Rizzo JD, Saber W, Hari PN. Bortezomib-based induction for transplant ineligible AL amyloidosis and feasibility of later transplantation. Bone Marrow Transplant. 2015 Jul;50(7):914-7. doi: 10.1038/bmt.2015.73. Epub 2015 Apr 27. PMID 25915809
- [Background] Gentile M, Vigna E, Recchia AG, Morabito L, Mendicino F, Giagnuolo G, Morabito F. Bendamustine in multiple myeloma. Eur J Haematol. 2015 Nov;95(5):377-88. doi: 10.1111/ejh.12609. Epub 2015 Jul 14. PMID 26085055
- [Background] Cheson BD, Rummel MJ. Bendamustine: rebirth of an old drug. J Clin Oncol. 2009 Mar 20;27(9):1492-501. doi: 10.1200/JCO.2008.18.7252. Epub 2009 Feb 17. PMID 19224851
- [Background] Flinn IW, van der Jagt R, Kahl BS, Wood P, Hawkins TE, Macdonald D, Hertzberg M, Kwan YL, Simpson D, Craig M, Kolibaba K, Issa S, Clementi R, Hallman DM, Munteanu M, Chen L, Burke JM. Randomized trial of bendamustine-rituximab or R-CHOP/R-CVP in first-line treatment of indolent NHL or MCL: the BRIGHT study. Blood. 2014 May 8;123(19):2944-52. doi: 10.1182/blood-2013-11-531327. Epub 2014 Mar 3. PMID 24591201
- [Background] Flinn IW, van der Jagt R, Kahl B, Wood P, Hawkins T, MacDonald D, Simpson D, Kolibaba K, Issa S, Chang J, Trotman J, Hallman D, Chen L, Burke JM. First-Line Treatment of Patients With Indolent Non-Hodgkin Lymphoma or Mantle-Cell Lymphoma With Bendamustine Plus Rituximab Versus R-CHOP or R-CVP: Results of the BRIGHT 5-Year Follow-Up Study. J Clin Oncol. 2019 Apr 20;37(12):984-991. doi: 10.1200/JCO.18.00605. Epub 2019 Feb 27. PMID 30811293
- [Background] Lentzsch S, Lagos GG, Comenzo RL, Zonder JA, Osman K, Pan S, Bhutani D, Pregja S, Sanchorawala V, Landau H. Bendamustine With Dexamethasone in Relapsed/Refractory Systemic Light-Chain Amyloidosis: Results of a Phase II Study. J Clin Oncol. 2020 May 1;38(13):1455-1462. doi: 10.1200/JCO.19.01721. Epub 2020 Feb 21. PMID 32083996
- [Background] Matsuda M, Gono T, Shimojima Y, Hoshii Y, Ikeda S. Phenotypic analysis of plasma cells in bone marrow using flow cytometry in AL amyloidosis. Amyloid. 2003 Jun;10(2):110-6. doi: 10.3109/13506120309041732. PMID 12964418
- [Background] Palladini G, Kastritis E, Maurer MS, Zonder J, Minnema MC, Wechalekar AD, Jaccard A, Lee HC, Bumma N, Kaufman JL, Medvedova E, Kovacsovics T, Rosenzweig M, Sanchorawala V, Qin X, Vasey SY, Weiss BM, Vermeulen J, Merlini G, Comenzo RL. Daratumumab plus CyBorD for patients with newly diagnosed AL amyloidosis: safety run-in results of ANDROMEDA. Blood. 2020 Jul 2;136(1):71-80. doi: 10.1182/blood.2019004460. PMID 32244252
- [Background] Jiang H, Acharya C, An G, Zhong M, Feng X, Wang L, Dasilva N, Song Z, Yang G, Adrian F, Qiu L, Richardson P, Munshi NC, Tai YT, Anderson KC. SAR650984 directly induces multiple myeloma cell death via lysosomal-associated and apoptotic pathways, which is further enhanced by pomalidomide. Leukemia. 2016 Feb;30(2):399-408. doi: 10.1038/leu.2015.240. Epub 2015 Sep 4. PMID 26338273
- [Background] Attal M, Richardson PG, Rajkumar SV, San-Miguel J, Beksac M, Spicka I, Leleu X, Schjesvold F, Moreau P, Dimopoulos MA, Huang JS, Minarik J, Cavo M, Prince HM, Mace S, Corzo KP, Campana F, Le-Guennec S, Dubin F, Anderson KC; ICARIA-MM study group. Isatuximab plus pomalidomide and low-dose dexamethasone versus pomalidomide and low-dose dexamethasone in patients with relapsed and refractory multiple myeloma (ICARIA-MM): a randomised, multicentre, open-label, phase 3 study. Lancet. 2019 Dec 7;394(10214):2096-2107. doi: 10.1016/S0140-6736(19)32556-5. Epub 2019 Nov 14. PMID 31735560
- [Background] Palladini G, Dispenzieri A, Gertz MA, Kumar S, Wechalekar A, Hawkins PN, Schonland S, Hegenbart U, Comenzo R, Kastritis E, Dimopoulos MA, Jaccard A, Klersy C, Merlini G. New criteria for response to treatment in immunoglobulin light chain amyloidosis based on free light chain measurement and cardiac biomarkers: impact on survival outcomes. J Clin Oncol. 2012 Dec 20;30(36):4541-9. doi: 10.1200/JCO.2011.37.7614. Epub 2012 Oct 22. PMID 23091105
- [Background] Palladini G, Hegenbart U, Milani P, Kimmich C, Foli A, Ho AD, Vidus Rosin M, Albertini R, Moratti R, Merlini G, Schonland S. A staging system for renal outcome and early markers of renal response to chemotherapy in AL amyloidosis. Blood. 2014 Oct 9;124(15):2325-32. doi: 10.1182/blood-2014-04-570010. Epub 2014 Aug 12. PMID 25115890
- [Background] Comenzo RL, Reece D, Palladini G, Seldin D, Sanchorawala V, Landau H, Falk R, Wells K, Solomon A, Wechalekar A, Zonder J, Dispenzieri A, Gertz M, Streicher H, Skinner M, Kyle RA, Merlini G. Consensus guidelines for the conduct and reporting of clinical trials in systemic light-chain amyloidosis. Leukemia. 2012 Nov;26(11):2317-25. doi: 10.1038/leu.2012.100. Epub 2012 Apr 5. PMID 22475872
- [Background] Staron A, Burks EJ, Lee JC, Sarosiek S, Sloan JM, Sanchorawala V. Assessment of minimal residual disease using multiparametric flow cytometry in patients with AL amyloidosis. Blood Adv. 2020 Mar 10;4(5):880-884. doi: 10.1182/bloodadvances.2019001331. PMID 32130406
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Background] Friedberg JW, Cohen P, Chen L, Robinson KS, Forero-Torres A, La Casce AS, Fayad LE, Bessudo A, Camacho ES, Williams ME, van der Jagt RH, Oliver JW, Cheson BD. Bendamustine in patients with rituximab-refractory indolent and transformed non-Hodgkin's lymphoma: results from a phase II multicenter, single-agent study. J Clin Oncol. 2008 Jan 10;26(2):204-10. doi: 10.1200/JCO.2007.12.5070. Erratum In: J Clin Oncol. 2008 Apr 10;26(11) 1911. PMID 18182663
- [Background] Kahl BS, Bartlett NL, Leonard JP, Chen L, Ganjoo K, Williams ME, Czuczman MS, Robinson KS, Joyce R, van der Jagt RH, Cheson BD. Bendamustine is effective therapy in patients with rituximab-refractory, indolent B-cell non-Hodgkin lymphoma: results from a Multicenter Study. Cancer. 2010 Jan 1;116(1):106-14. doi: 10.1002/cncr.24714. PMID 19890959
- [Background] Fischer K, Cramer P, Busch R, Stilgenbauer S, Bahlo J, Schweighofer CD, Bottcher S, Staib P, Kiehl M, Eckart MJ, Kranz G, Goede V, Elter T, Buhler A, Winkler D, Kneba M, Dohner H, Eichhorst BF, Hallek M, Wendtner CM. Bendamustine combined with rituximab in patients with relapsed and/or refractory chronic lymphocytic leukemia: a multicenter phase II trial of the German Chronic Lymphocytic Leukemia Study Group. J Clin Oncol. 2011 Sep 10;29(26):3559-66. doi: 10.1200/JCO.2010.33.8061. Epub 2011 Aug 15. PMID 21844497
- [Background] Martin T, Strickland S, Glenn M, Charpentier E, Guillemin H, Hsu K, Mikhael J. Phase I trial of isatuximab monotherapy in the treatment of refractory multiple myeloma. Blood Cancer J. 2019 Mar 29;9(4):41. doi: 10.1038/s41408-019-0198-4. PMID 30926770
- [Background] Munshi NC, Avet-Loiseau H, Rawstron AC, Owen RG, Child JA, Thakurta A, Sherrington P, Samur MK, Georgieva A, Anderson KC, Gregory WM. Association of Minimal Residual Disease With Superior Survival Outcomes in Patients With Multiple Myeloma: A Meta-analysis. JAMA Oncol. 2017 Jan 1;3(1):28-35. doi: 10.1001/jamaoncol.2016.3160. PMID 27632282
- [Background] Laabi Y, Gras MP, Carbonnel F, Brouet JC, Berger R, Larsen CJ, Tsapis A. A new gene, BCM, on chromosome 16 is fused to the interleukin 2 gene by a t(4;16)(q26;p13) translocation in a malignant T cell lymphoma. EMBO J. 1992 Nov;11(11):3897-904. doi: 10.1002/j.1460-2075.1992.tb05482.x. PMID 1396583
- [Background] Novak AJ, Darce JR, Arendt BK, Harder B, Henderson K, Kindsvogel W, Gross JA, Greipp PR, Jelinek DF. Expression of BCMA, TACI, and BAFF-R in multiple myeloma: a mechanism for growth and survival. Blood. 2004 Jan 15;103(2):689-94. doi: 10.1182/blood-2003-06-2043. Epub 2003 Sep 25. PMID 14512299
- [Background] Thompson JS, Schneider P, Kalled SL, Wang L, Lefevre EA, Cachero TG, MacKay F, Bixler SA, Zafari M, Liu ZY, Woodcock SA, Qian F, Batten M, Madry C, Richard Y, Benjamin CD, Browning JL, Tsapis A, Tschopp J, Ambrose C. BAFF binds to the tumor necrosis factor receptor-like molecule B cell maturation antigen and is important for maintaining the peripheral B cell population. J Exp Med. 2000 Jul 3;192(1):129-35. doi: 10.1084/jem.192.1.129. PMID 10880534
- [Background] Coquery CM, Erickson LD. Regulatory roles of the tumor necrosis factor receptor BCMA. Crit Rev Immunol. 2012;32(4):287-305. doi: 10.1615/critrevimmunol.v32.i4.10. PMID 23237506
- [Background] O'Connor BP, Raman VS, Erickson LD, Cook WJ, Weaver LK, Ahonen C, Lin LL, Mantchev GT, Bram RJ, Noelle RJ. BCMA is essential for the survival of long-lived bone marrow plasma cells. J Exp Med. 2004 Jan 5;199(1):91-8. doi: 10.1084/jem.20031330. PMID 14707116
- [Background] Xu S, Lam KP. B-cell maturation protein, which binds the tumor necrosis factor family members BAFF and APRIL, is dispensable for humoral immune responses. Mol Cell Biol. 2001 Jun;21(12):4067-74. doi: 10.1128/MCB.21.12.4067-4074.2001. PMID 11359913
- [Background] Laurent SA, Hoffmann FS, Kuhn PH, Cheng Q, Chu Y, Schmidt-Supprian M, Hauck SM, Schuh E, Krumbholz M, Rubsamen H, Wanngren J, Khademi M, Olsson T, Alexander T, Hiepe F, Pfister HW, Weber F, Jenne D, Wekerle H, Hohlfeld R, Lichtenthaler SF, Meinl E. gamma-Secretase directly sheds the survival receptor BCMA from plasma cells. Nat Commun. 2015 Jun 11;6:7333. doi: 10.1038/ncomms8333. PMID 26065893
- [Background] Sanchez E, Li M, Kitto A, Li J, Wang CS, Kirk DT, Yellin O, Nichols CM, Dreyer MP, Ahles CP, Robinson A, Madden E, Waterman GN, Swift RA, Bonavida B, Boccia R, Vescio RA, Crowley J, Chen H, Berenson JR. Serum B-cell maturation antigen is elevated in multiple myeloma and correlates with disease status and survival. Br J Haematol. 2012 Sep;158(6):727-38. doi: 10.1111/j.1365-2141.2012.09241.x. Epub 2012 Jul 18. PMID 22804669
- [Background] Godara A, Zhou P, Kugelmass A, Ma X, Rosenthal B, Toskic D, Fogaren T, Varga C, Comenzo RL. Presence of soluble and cell-surface B-cell maturation antigen in systemic light-chain amyloidosis and its modulation by gamma-secretase inhibition. Am J Hematol. 2020 May;95(5):E110-E113. doi: 10.1002/ajh.25734. Epub 2020 Jan 29. No abstract available. PMID 31951032
- [Background] Dispenzieri A, Gertz MA, Kyle RA, Lacy MQ, Burritt MF, Therneau TM, Greipp PR, Witzig TE, Lust JA, Rajkumar SV, Fonseca R, Zeldenrust SR, McGregor CG, Jaffe AS. Serum cardiac troponins and N-terminal pro-brain natriuretic peptide: a staging system for primary systemic amyloidosis. J Clin Oncol. 2004 Sep 15;22(18):3751-7. doi: 10.1200/JCO.2004.03.029. PMID 15365071
- [Background] Wechalekar AD, Schonland SO, Kastritis E, Gillmore JD, Dimopoulos MA, Lane T, Foli A, Foard D, Milani P, Rannigan L, Hegenbart U, Hawkins PN, Merlini G, Palladini G. A European collaborative study of treatment outcomes in 346 patients with cardiac stage III AL amyloidosis. Blood. 2013 Apr 25;121(17):3420-7. doi: 10.1182/blood-2012-12-473066. Epub 2013 Mar 11. PMID 23479568
- See also: Teva Pharmaceuticals International (bendamustine hydrochloride) [package insert] — https://www.accessdata.fda.gov/drugsatfda_docs/label/2015/208194s000lbl.pdf
- See also: Sanofi Aventis US. Sarclisa (isatuximab-irfc) [package insert]. — https://www.accessdata.fda.gov/drugsatfda_docs/label/2020/761113s000lbl.pdf